CLINICAL TRIAL: NCT01651923
Title: PHARMACODYNAMICS ASSESSMENT PRODUCT HEPARIN SODIUM (INTRAVENOUSLY) OF THE SWINE 5.000UI/ML OF BLAU FARMACÊUTICA S/A IN HEALTHY SUBJECTS IN COMPARISON OF SODIUM HEPARIN APP PHARMACEUTICALS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HEPBLA0312IV-I; Versão 01 - 15/03/2012
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: subjects
MeSH Terms: interventions — Heparin

ARMS (2):
- Group A (Other): First periody: Heparin Test Drug (Blau Farmacêutica S/A)
  Secundy periody: Heparin Comparator Drug (APP Pharmaceuticals)
  Interventions: Drug: Heparin
- Group B (Other): First periody: Heparin Comparator Drug (APP Pharmaceuticals)
  Secundy periody: Heperin Test Drug (Blau Farmacêutica S/A)
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Heparin — Whereas it will be a crossover study with two periods, each drug will be administered only once, at a dose of 5.000UI. In each period, the drug will be administered intravenously.
  Other Names: Sodium heparin (Blau Farmacêutica S/A); Sodium heparin (App Pharmaceuticals)

SUMMARY:
The objective of this clinical, randomized, crossover, is to assess the pharmacodynamic profile of the drug Heparin Sodium from swine (intravenously), manufactured and marketed by Laboratory Blau Farmacêutica S/A, compared to the product of Heparin Sodium ® company APP Pharmaceuticals, through the determination of activity of the following markers:

* Anti-FXa;
* Anti-FIIA.

DETAILED DESCRIPTION:
The pharmacodynamic profile of the drug will be assessed through:

* Reason for Anti-FXa activity / Anti-FIIA;
* TFPI activity.

The aPTT activity marker will be evaluated as an exploratory objective.

ELIGIBILITY:
Inclusion Criteria:

* a) Confirm the voluntary participation and agree to all the purposes of the study by signing and dating the IC in two ways; b) Being male, aged between 18 and 55 years old and clinically healthy; c) BMI ≥ 18.5 and ≤ 30.

Exclusion Criteria:

* a) Participation in clinical trials in the 12 months preceding the survey; b) Presence of pulmonary diseases, cardiovascular, neurological, endocrine, gastrointestinal, genitourinary or other systems; c) acute illness in the period up to 07 days before the beginning of the study; d) determining Chronic administration of medications, such as hypertension, diabetes or any other that requires continued use of any drug; e) Hemoglobin <13 g / dL; f) Continuous use of oral anticoagulants, platelet inhibitors or anti-inflammatory; g) Use of medications that interact with heparin (see Section 7.8.1); h) history of gastrointestinal bleeding, deep vein thrombosis or pulmonary embolism; i) History of coagulopathy and bleeding diathesis; j) Presence of bruises on physical examination. k) Changes in skin or subcutaneous tissue of the place where the injection is made (eg liposuction in the abdomen).

  l) absolute platelet count below 100 x 109 / L; m) A history of acute haemorrhage in the last 30 days; n) history of sensitivity to biological products derived from mammalian albumin or any component of the formulation;

  a) history of allergy or major disease Steven Johnson; p) History of present use or there are at least 12 months of tobacco; q) current or previous history (less than 12 months) of illicit drug use;

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamic of activity of markers: Anti-Fxa and Anti-FIIA | 0:20, 0:10 before administration and 0:10, 0:20, 0:30, 0:45, 1, 1:30, 2, 2:30, 3, 3:30, 4, 4:30 , 5, 6, 8, 12 and 24 hours after drug administration.
  Blood samples

SECONDARY OUTCOMES:
Pharmacodynamic of the ratio between the activity Anti-FXa/Anti-FIIa and the activity of TFPI and TTPa | TFPI: 0:20, 0:10 before administration and 0:10, 0:20, 0:30, 0:45, 1, 1:30, 2, 2:30, 3, 3:30, 4, 4:30 , 5, 6, 8, 12 and 24 hours after drug administration. TTPa: 0:20, 0:10 before administration and 1 h, 4h, 8h, 12h and 24h after drug administration
  Blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clínica Pesquisa e Desenvolvimento Ltda., Valinhos, São Paulo, Brazil